CLINICAL TRIAL: NCT04833907
Title: Phase 1/2, Open Label, Sequential Cohort Study of a Single Intracranial Dose of AVASPA Gene Therapy for Treatment of Children With Typical Canavan Disease
Brief Title: rAAV-Olig001-ASPA Gene Therapy for Treatment of Children With Typical Canavan Disease
Acronym: CAN-GT
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Myrtelle Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-GT
Record Dates: First submitted 2021-03-24; First posted 2021-04-06 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-01

CONDITIONS: Canavan Disease
Keywords: Canavan Disease; Gene Therapy; Aspartoacylase; N-Acetyl-Aspartate; Oligodendrocyte; Leukodystrophy; Adeno-Associated Virus Vector; Autosomal Recessive Disorder; Neurodegenerative; White Matter Disorder
MeSH Terms: conditions — Canavan Disease | interventions — Levetiracetam; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3.7 x 10^13 v.g. rAAV-Olig001-ASPA (Experimental): 3.7 x 10^13 v.g. of rAAV-Olig001-ASPA administered as a single dose neurosurgically to the brain via 2 pre-defined intracerebroventricular sites
  Interventions: Drug: rAAV-Olig001-ASPA; Drug: Levetiracetam; Drug: Prednisone

INTERVENTIONS:
Drug: rAAV-Olig001-ASPA — Intracerebroventricular administration of a single dose
  Other Names: MYR-101
Drug: Levetiracetam — Keppra daily dose (20-50 mg/kg/day divided twice daily administered orally or per G-tube) in the post-operative period and continued for 3 months per standard of care to prevent seizure activity.
  Other Names: Keppra
Drug: Prednisone — Post-operatively, a 3-month steroid taper is planned to prevent or reduce possible delayed immunological responses. This tapering regimen will consist of 0.5 mg/kg/day prednisone during weeks 1-4; followed by 0.3 mg/kg/day prednisone during weeks 5-8; and 0.1mg prednisone during weeks 9-12, then off. If there is evidence of new inflammation on MRI at 3-months on T2 FLAIR, the steroid taper will be extended for an additional 3 months or we will transition to steroid-sparing immunosuppression.

SUMMARY:
Canavan Disease is a congenital white matter disorder caused by mutations to the gene encoding for aspartoacylase (ASPA). Expression of ASPA is restricted to oligodendrocytes, the sole white matter producing lineage in the brain. ASPA supports myelination in the capacity of its sole known function, namely, the catabolism of N-acetylaspartate (NAA). Inherited mutations that result in loss of ASPA catabolic activity result in a typically severe phenotype of Canavan Disease, characterized by chronically elevated brain NAA, gross motor abnormalities, hypomyelination, progressive spongiform degeneration of the brain, epilepsy, blindness, and a short life expectancy. Disease severity is correlated with residual levels of enzyme activity. Reconstitution of ASPA function in oligodendrocytes of the brains of Canavan patients is expected to rescue NAA metabolism in its natural cellular compartment and support myelination/remyelination by resident white matter producing cells. This protocol directly targets oligodendrocytes in the brain, which are intimately involved with disease initiation and progression. Targeting oligodendrocytes offers the safest and most direct therapy for affected individuals.

The latest generation AAV viral vector (rAAV-Olig001-ASPA) will be administered to patients using neurosurgical procedure which involves direct administration of gene therapy to affected regions of the brain. Outcome measures for the open label clinical trial include longitudinal clinical assessments and brain imaging.

Currently, there is no effective treatment for Canavan Disease. The purpose of this study is to validate a new technology targeted to the cells most affected by Canavan Disease in the safest way possible.

The study investigators are committed to supporting the Rare Disease & Canavan Disease Communities. For more information, please contact Jordana Holovach, Head of Communications and Community at PatientAdvocacy@myrtellegtx.com.

DETAILED DESCRIPTION:
rAAV-Olig001-ASPA is the first gene therapy designed to target the oligodendrocytes, which are critical for myelination and brain development.

This study is a Phase 1/2 First-In-Human protocol designed to obtain safety, pharmacodynamics, and efficacy data following neurosurgical administration of a single dose of rAAV-Olig001-ASPA delivered intracerebroventricularly in up to 24 children with Canavan Disease.

Patients with a diagnosis of typical Canavan Disease who meet all eligibility criteria may be enrolled in this open-label, sequential cohort study of a single dose of rAAV-Olig001-ASPA.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of typical CD by a board certified neurologist.
* Written informed consent from parent(s)/guardian(s). Consent to enroll into the study will include a written agreement to comply with all the conditions of the study, including attendance at follow-up visits.
* For cohort 1: age more than 36 months and up to 60 months.
* For cohort 2: age between 15 months and 36 months.
* For cohort 3: age less than 15 months.

Exclusion Criteria:

* At the discretion of the PI, any significant chronic medical condition, including, but not limited to neurological, cardiac, hepatic, renal, hematological, gastrointestinal, endocrine, pulmonary, or infectious disease, which would put the subject at increased risk during surgery or which would interfere with participation in the study, interpretation of safety monitoring, or the integrity of the study data.
* History of severe allergic reaction or anaphylaxis.
* Past participation in gene therapy trials or receipt of any other investigational product within 6 months prior to enrollment.
* Prior intracranial surgery.
* Any absolute contraindication to immunosuppression.
* Any absolute contraindication to MRI.
* Any vaccination less than 1 month prior to gene therapy.
* Anticipated life expectancy of less than 12 months for any reason.
* GMFM-88 total raw score >35%.
* Clinically significant out-of-range lab values, at the discretion of clinical PI.

Ages: 3 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | 12 Months Post Dose
  Number, severity, and causal relationship of any adverse event (to either the gene therapy and/or surgical trial procedures required for vector administration) using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Myelination | 12 Months Post Dose
  Change from baseline measured by cerebral Synthetic Magnetic Resonance Imaging (SyMRI)
N-Acetyl-Aspartate (NAA) concentrations in the Brain | 12 Months Post Dose
  N-Acetyl-Aspartate concentrations will be assessed with nuclear Magnetic Resonance Spectroscopy (nMRS) between pre- and post-treatment and as compared to historical controls.
Neurological Evaluation - Motor Function | 12 Months Post Dose
  Motor Function will be analyzed using the Gross Motor Function Measure (GMFM)-88 scale for motor function assessment before and after vector administration and compared to historical controls. The GMFM consists of 5 scales: Lying and Rolling, Sitting, Crawling and Kneeling, Standing and Walking, Running and Jumping. The total scores range from 0 to 264. The lower the score on GMFM, the weaker the ability; the higher the score, the greater the ability.
Neurological Evaluation - Neurocognitive Function | 12 Months Post Dose
  Neurocognitive function will be assessed using the Mullen Scales of Early Learning (MSEL) before and after vector administration and compared to historical controls. The MSEL is a cognitive test to measure cognitive ability and language development. The MSEL test has five scales: Gross motor, Visual reception, Fine motor, Receptive language, and Expressive language. The total scores range from 0 to 197. The lower the score on MSEL, the weaker the ability; the higher the score, the greater the ability.
Neurological Evaluation - Spasticity | 12 Months Post Dose
  Will be assessed using the Canavan Neurological Evaluation before and after vector administration and compared to historical controls.
Seizure Assessment | 12 Months Post Dose
  Will be assessed based on reported seizure activity and Electroencephalograms alpha, beta, delta, and theta wave frequencies (Hz).
NAA concentration measured in Cerebrospinal Fluid (CSF) | 6 months
  CSF will be collected via lumbar puncture and analyzed to assess concentrations of N-Acetyl-Aspartate.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lober, MD, PhD, Principal Investigator — Dayton Children's Hospital
Locations (1):
- Dayton Children's Hospital, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Francis JS, Markov V, Wojtas ID, Gray S, McCown T, Samulski RJ, Figueroa M, Leone P. Preclinical biodistribution, tropism, and efficacy of oligotropic AAV/Olig001 in a mouse model of congenital white matter disease. Mol Ther Methods Clin Dev. 2021 Jan 21;20:520-534. doi: 10.1016/j.omtm.2021.01.009. eCollection 2021 Mar 12. PMID 33614826
- [Background] Francis JS, Wojtas I, Markov V, Gray SJ, McCown TJ, Samulski RJ, Bilaniuk LT, Wang DJ, De Vivo DC, Janson CG, Leone P. N-acetylaspartate supports the energetic demands of developmental myelination via oligodendroglial aspartoacylase. Neurobiol Dis. 2016 Dec;96:323-334. doi: 10.1016/j.nbd.2016.10.001. Epub 2016 Oct 4. PMID 27717881
- [Derived] Leone P, Lober RM, Francis J, Flamini O, Cecil KM, Shera D, Janson CG. Oligodendrocyte-targeted adeno-associated virus gene therapy for Canavan disease in children: a phase 1/2 trial. Nat Med. 2025 Nov;31(11):3772-3779. doi: 10.1038/s41591-025-03919-w. Epub 2025 Sep 16. PMID 40957959
- See also: Canavan Disease — https://rarediseases.info.nih.gov/diseases/5984/canavan-disease
- See also: Canavan Disease Research — https://research.rowan.edu/research-areas/biomedical/leone/index.html
- See also: Canavan Disease Advocacy, Research, Patient assistance, Education — https://curecanavanfund.org
- See also: Canavan Disease Advocacy, Research, Patient assistance, Education — http://www.canavan.org
- See also: Canavan Disease Advocacy, Research, Patient assistance, Education — https://www.canavanfoundation.org
- See also: Canavan Disease Advocacy, Research, Patient assistance, Education — https://www.canavanresearch.org
- See also: Canavan Disease Advocacy, Research, Patient assistance, Education — https://www.ntsad.org